CLINICAL TRIAL: NCT00712023
Title: Effect of Forced-air Warming and Circulating-water Mattress in Preventing Heat Loss During Vascular Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: SUWANNEE SURASERANIVONGSE, Department of Anesthesiology, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Si 196/2007; 003(1)/50
Record Dates: First submitted 2008-05-14; First posted 2008-07-09 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2008-04

CONDITIONS: Hypothermia; Vascular Surgery; Forced-air Warming Mattress; Circulating-water Mattress
Keywords: Hypothermia; Vascular surgery; Forced-air warming mattress; Circulating-water mattress
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): warming by circulating-water mattress
  Interventions: Device: warming device (a reusable, custom-made forced- air warming mattress)
- 2 (No Intervention): Forced-air warming mattress

INTERVENTIONS:
Device: warming device (a reusable, custom-made forced- air warming mattress) — 2=forced-air warming mattress
  1=circulating-water mattress
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether a custom-made forced-air warming mattress can prevent heat loss in patients undergoing vascular surgery better than a circulating-water mattress

DETAILED DESCRIPTION:
A reusable, custom-made forced-air warming mattress was made of a light to medium weight water resistant canvas, sewn like mattress with 2 arms placed underneath the patient. An open hole at proximal part of one arm was designed to attach with a hose of warm air delivery device. Small holes (2-3 mm2), 5 inches apart were punched on the upper surface of this mattress around the patient except for the area underneath the patient that the holes were 9 inches apart. The weight of the patient will obstruct the air flow and prevent direct blowing of warm air onto the underside of patients. There is a special appendage connected to the upper part of mattress which can connect warm air to cover the patient's chest. There is a special appendage connected to the upper part of mattress which can convect warm air to cover the patient's chest. The mattress is 97 inches x 97 inches, with 2 arms of 25 inches x 16 inches and a special appendage of 45 inches x 12 inches for covering the chest with warm air delivery. This size is proper for patient of 170 cm. height. In order to reuse it, the mattress can be washed, dried and sterilized by gas or autoclaved for more than 50 times. A sterile sheet well enhance the sterile environment of the operating field.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing vascular surgery

Exclusion Criteria:

Preoperative fever

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
skin and nasopharyngeal temperature | 180 min

SECONDARY OUTCOMES:
burn wound | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Suwannee Suraseraniwongse, MD, Principal Investigator — Mahidol University
Locations (1):
- Departnment of Anesthesiology,Siriraj Hospital, Mahidol University, Bangkok, Thailand